CLINICAL TRIAL: NCT04565106
Title: Automatic Oxygen Titration With O2matic® to Patients Admitted With COVID-19 and Hypoxemic Respiratory Failure
Acronym: O2matic-COVI
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Ejvind Frausing Hansen, Chief Physician, Hvidovre University Hospital
Other Study IDs: O2matic-COVID
Record Dates: First submitted 2020-09-24; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Hypoxemic Respiratory Failure; Hypoxemia
Keywords: O2matic; Closed-loop
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Closed-loop control of oxygen supplementation by O2matic — Closed-loop control of oxygen supplementation to achieve a target SpO2 of 92 - 96 %

SUMMARY:
Patients with coronavirus disease (COVID-19) and pneumonitis often have hypoxemic respiratory failure and a need of supplementary oxygen. Guidelines recommend controlled oxygen, for most patients with a recommended interval of SpO2 between 92 and 96 %. We aimed to determine if closed-loop control of oxygen was feasible in patients with COVID-19 and could maintain SpO2 in the specified interval.

DETAILED DESCRIPTION:
Patients with coronavirus disease (COVID-19) and pneumonitis often have hypoxemic respiratory failure and a need of supplementary oxygen. Guidelines recommend controlled oxygen, for most patients with a recommended interval of SpO2 between 92 and 96 %. We aimed to determine if closed-loop control of oxygen was feasible in patients with COVID-19 and could maintain SpO2 in the specified interval.

Patients were prospectively enrolled in an observational study on a medical ward dedicated to patients with COVID-19. Closed-loop controlled oxygen was delivered by O2matic® which can deliver 0-15 liters/min and adjusts flow every second based on 15 seconds averaging of SpO2 measured by pulse oximetry. Lung function parameters were measured at admission.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Positive COVID-19 PCR analysis in pharyngeal swab or in tracheal secretion
* Need oxygen supply to maintain SpO2 ≥ 92 %
* Able to comply with continuous measurement of SpO2 by pulse oximetry.

Exclusion Criteria:

* Need of oxygen supply > 10 liters/min at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with COVID-19 pneumonitis and in need of oxygen supplementation
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Time in SpO2 target | 1 week
  Time in SpO2 target of 92-96 %

SECONDARY OUTCOMES:
Time with SpO2 not more than 2 % outside target | 1 week
  Time with SpO2 not more than 2 % outside target
Time with SpO2 more than 2 % outside target | 1 week
  Time with SpO2 more than 2 % outside target
Time with SpO2 < 85 % | 1 week
  Time with SpO2 < 85 %

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, PhD, Study Chair — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No